CLINICAL TRIAL: NCT06545578
Title: Effect of Motor Control Exercise Combined With Laser Or TENS on Pain, Range of Motion, and Functional Disability on Obese Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Ababa, lecturer of internal physical therapy, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T-ORTH-05/2023-511
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Back Pain; Obesity; Motor Control Exercises; Laser Therapy
MeSH Terms: conditions — Back Pain; Obesity | interventions — Low-Level Light Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A): (Experimental): Group A received motor control exercises with low level laser therapy
  Interventions: Other: low-level laser therapy; Other: motor control exercises
- Group (B): (Experimental): Group B received motor control exercises with transcutaneous electrical nerve stimulation
  Interventions: Other: TENS; Other: motor control exercises

INTERVENTIONS:
Other: low-level laser therapy — The Low-level laser (LLL) pain-relief instrument RG-300IB (code E22), manufactured in China, was utilized for low-level laser therapy (LLLT) in Group A . The therapy employed a wavelength of 830 nm (near infrared) and involved careful skin contact hygiene at specified positions, 2.5 and 3.5 cm laterally from the spinous process (L4, L5, or S1) and one distal level segment. The laser operated at a repetition rate of 5,000, with a power density of 300 mW/cm2 and a power output of 10 mW. Each point received 3 J of energy, resulting in a density of 3 J/cm2, with four points. The spot size was 1 cm, and each point received a 30-second treatment. The energy was administered three times per week for four weeks
  Arms: Group (A):
Other: TENS — TENS Intelect Advanced device (Chattanooga, Mouguerre, France). The parameters for TENS stimulation included a frequency range of 60-80 Hz, a pulse width of 50-80 ms, and an intensity of 10-30 mA. Before commencing therapy, patients were provided information regarding the therapeutic approach and any potential adverse effects. During the procedure, two channels (four electrodes) were employed, with one set placed on the right and one on the left paraspinal muscles at the level of L2-L4. Active electrodes from the other channels were affixed 1.5 cm laterally to the spine, while passive electrodes were positioned 3 cm away. TENS therapy was utilized for 30 minutes in Group B, and the intensity of the pain and discomfort was adjusted to the patient's tolerance level.
  Arms: Group (B):
Other: motor control exercises — Training in coordinated trunk muscle action, including decreasing overactive superficial muscles and independent activation of deep muscles (such as transversus abdominis and multifidus). Exercises for the pelvic floor muscles, controlling respiration, and regulating the position and movement of the spine were added to these exercises.

SUMMARY:
This randomized study aimed to assess the impact of MCE in conjunction with LLLT and MCE in conjunction with TENS on pain levels, ROM, and functional disability in obese patients with LBP.

DETAILED DESCRIPTION:
Sixty obese male and female patients with LBP participated in this study. After providing informed consent, they were randomly divided into two equal groups, with Group A receiving MCE combined with LLLT and Group B receiving MCE combined with TENS.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were the following:

* patients aged 40 to 77 years
* non-athletic, have a BMI > 25
* complaining of LBP.

Exclusion Criteria:

The exclusion criteria were the following:

* vertebral fractures
* surgical spinal fixation
* rheumatic disorders
* any underlying medical condition that may be causing back pain, including:
* malignancy
* viscerogenic causes
* infection, systemic disease of the muscles and skeletal system,
* sensory dysfunction
* neuromuscular diseases like multiple sclerosis.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-06 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
The pain was evaluated utilizing the visual analog scale (VAS) | before treatment and 4 weeks after treatment
  It comprises a 10-centimeter-long horizontal line secured at both ends with anchors. The initial anchor signifies the absence of pain, whereas the final anchor represents the most terrible pain. The patient was instructed to indicate the point through the line that most accurately represented the intensity of discomfort. The measurement was obtained by tracing the distance from the zero extremities to the patient's mark
the functional disability, the Oswestry disability questionnaire version 2.0 | before treatment and 4 weeks after treatment
  Assessing functional disability in patients afflicted with LBP is accomplished with a valid and dependable instrument. There are six possible responses to each of the ten queries, which includes the daily functional disability. The patient chose the response that best described his impairment. Scores up to 50 are possible and are divided as follows: each question takes 5, the first statement takes 0, and the sixth statement takes 5 scores. The maximum score in this study was 45. All scores were subsequently tallied and converted to a percentage of the total score. A greater score is indicative of a severe disability. Scores between 0 and 20 represent minimal disability. Disability levels are classified as follows: scores between 40 and 60 indicate moderate disability; scores between 60 and 80 indicate disabled disability; and scores between 80 and 100 indicate bedridden patients
1- Assessment of lumbar flexion ROM | before treatment and 4 weeks after treatment
  The researcher positioned himself behind the patient standing to use his thumbs to identify the two posterior superior iliac spines (PSIS). He then delineated these two spines with a line on the skin, with the first mark located at the midpoint of the line and the second mark positioned 15 cm above. Subsequently, the researcher directed the patient to flex forward to the greatest extent possible while remaining within the boundaries of pain
2- Assessment of lumbar extension ROM | before treatment and 4 weeks after treatment
  Instructing the patient to bend backward to the best of his ability within the boundaries of pain, the investigator established a line on the skin and positioned himself behind the standing patient to distinguish between the two PSIS with his thumbs. The first mark was located at the midpoint of this line, and the second mark was positioned 15 cm above the first.
3- Assessment of lumbar side bending ROM | before treatment and 4 weeks after treatment
  As the patient assumed an erect position with heels, buttocks, and shoulders against the wall and a lateral bend without elevating the opposing foot off the ground, the investigator determined the distance between the third fingertip and the floor.

CONTACTS AND LOCATIONS:
Locations (1):
- Ababa physical therapy center, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No